CLINICAL TRIAL: NCT03042494
Title: Effect of Prebiotic Intake on Gut Microbiota in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: General Mills (Industry)
Responsible Party: Principal Investigator, Dr. Raylene Reimer, Professor, University of Calgary
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: REB16-0388
Record Dates: First submitted 2017-02-01; First posted 2017-02-03 (Estimated); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Healthy
Keywords: Prebiotic; Gut microbiota; Dietary fiber; Gastrointestinal tolerance
MeSH Terms: interventions — Prebiotics

STUDY DESIGN:
Intervention Model Description: Crossover design with 4 week washout period.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): Isocaloric food without the test prebiotic.
  Interventions: Dietary Supplement: Control
- Prebiotic (Experimental): Prebiotic consumed as one daily serving of 7 g in Group 1 and consumed as one daily serving of 2.5-3 g in Group 2.
  Interventions: Dietary Supplement: Prebiotic

INTERVENTIONS:
Dietary Supplement: Control — Isocaloric food without the test prebiotic.
  Arms: Control
Dietary Supplement: Prebiotic — Prebiotic consumed as 7 g/d in a snack food in Group 1 and consumed as 2.5-3 g/d in a snack food in Group 2.
  Arms: Prebiotic

SUMMARY:
In recent years, the importance of the gut microbiota to human health has been demonstrated. In adulthood, the microbial profile is relatively stable, yet can be transiently altered by factors such as diet or antibiotic treatment. Such changes may be beneficial, as gut microbiota has been shown to differ in normal versus disease states including inflammatory bowel disease, obesity, type 2 diabetes and fatty liver disease. Given this relationship, there is intense interest in designing interventions that positively influence the gut microbial profile. Prebiotics are non-digestible, fermentable oligo- and polysaccharides that alter the colonic environment in favour of health-promoting bacterial species, such as bifidobacteria which selectively ferment prebiotics. Given the ability of prebiotics to beneficially alter the microbial profile, there is a need to identify the dosing requirements to positively modulate the gut microbiota. This study will test the effect of two doses of prebiotic on gut microbiota taxonomy and diversity.

DETAILED DESCRIPTION:
The primary objective is to determine the effect of 4 week intake of a moderate dose (7 g/d) or low dose (2.5-3 g/d) of prebiotic on gut microbiota profiles in healthy adults compared to a non-prebiotic containing control.

The primary outcome is change in microbial composition (measured via 16S rRNA sequencing).

The secondary outcomes are change in gastrointestinal (GI) tolerance (measured via questionnaire); change in fecal short chain fatty acids; and change in quality of life.

This study will consist of two separate trials of 12 week duration. Each trial will be performed in a double-blind, randomized, placebo-controlled crossover manner with a 4 week intervention period followed by a 4 week wash-out period and final 4 week cross over.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects who are regular snack consumers
* Not obese (BMI ≥ 18.5 kg/m2 and ≤ 29.9 kg/m2)
* 18 and 65 years of age
* Stable bodyweight for at least 3-months prior to the study.

Exclusion Criteria:

* Chronic disease including but not limited to type 1 or 2 diabetes, cardiovascular disease, liver or pancreas disease.
* Major gastrointestinal surgery
* Pregnant or lactating
* Antibiotic use in the preceding 3 months
* Currently consume probiotic or prebiotics supplements
* Currently consume more than 15 g/d of fiber in women and 18 g/d in men
* Are following a diet or exercise regime designed for weight loss
* Have a BMI greater than 29.9 kg/m2.
* Subjects who are required to start an antibiotic regime during the study will be withdrawn.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-05-15 (Actual); Primary Completion 2017-05-25 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in baseline fecal bifidobacteria at 4 weeks | 4 weeks in cross-over design
  Assessed with 16S rRNA sequencing.

SECONDARY OUTCOMES:
Change in baseline fecal short chain fatty acid concentrations at 4 weeks | 4 weeks in cross-over design
  Analyzed with gas chromatography/mass spectrophotometry
Change in baseline gastrointestinal tolerance at 4 weeks | 4 weeks in cross-over design
  Analyzed with questionnaire
Change in baseline quality of life rating at 4 weeks | 4 weeks in cross-over design
  Measured with SF-36 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Raylene Reimer, PhD, RD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reimer RA, Soto-Vaca A, Nicolucci AC, Mayengbam S, Park H, Madsen KL, Menon R, Vaughan EE. Effect of chicory inulin-type fructan-containing snack bars on the human gut microbiota in low dietary fiber consumers in a randomized crossover trial. Am J Clin Nutr. 2020 Jun 1;111(6):1286-1296. doi: 10.1093/ajcn/nqaa074. PMID 32320024